CLINICAL TRIAL: NCT06616571
Title: A Randomized, Open-label, Interventional, Real-world Study to Compare the Efficacy and Safety of QL0605 Administered at Different Timepoints After Chemotherapy.
Brief Title: Compare the Efficacy and Safety of QL0605 Injections at Different Timepoints
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QL0605-401
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Chemotherapy-Induced Febrile Neutropenia
Keywords: Febrile Neutropenia, Breast Cancer, Chemotherapy
MeSH Terms: conditions — Chemotherapy-Induced Febrile Neutropenia; Febrile Neutropenia; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24h group (Experimental)
  Interventions: Drug: QL0605(PEG-rhG-CSF)
- 48h group (Active Comparator)
  Interventions: Drug: QL0605(PEG-rhG-CSF)

INTERVENTIONS:
Drug: QL0605(PEG-rhG-CSF) — Eligible patients are scheduled to receive 2 cycles of chemotherapy every three weeks. During each chemotherapy cycle QL0605 is injected 24 hours s.c. post chemotherapy application.
Drug: QL0605(PEG-rhG-CSF) — Eligible patients are scheduled to receive 2 cycles of chemotherapy every three weeks. During each chemotherapy cycle QL0605 is injected 48 hours s.c. post chemotherapy application.

SUMMARY:
The goal of this real-world study is to compare the efficacy and safety of QL0605 administered 24 hours and 48 hours after chemotherapy in breast cancer patients.

DETAILED DESCRIPTION:
Patients with stage invasive breast cancer who were scheduled to receive at least 2 cycles of adjuvant or neoadjuvant chemotherapy with TAC/TC/TCbH regimen were eligible for this multicenter, open-label, randomized trial. Patients were randomized (2:1) to receive QL0605 24 hours (24h group) or 48 hours (48h group) after the end of each cycle of chemotherapy. The primary endpoint was the incidence rate of FN for cycle 1. The secondary endpoints included the incidence rates of grade 3/4 neutropenia, chemotherapy dose reduction and chemotherapy delay due to neutropenia, antibiotic administration, the pain (bone, muscle, or joint), ect.

ELIGIBILITY:
Inclusion Criteria:

* Aged≥18 years；
* The expected survival period is more than 3 months;
* ECOG≤ 2;
* Invasive breast cancer diagnosed by histopathology;
* Plan to receive TAC, TC or TCbH chemotherapy;
* Subjects with good hematology, liver, lung and kidney function ;
* Signed informed consent.

Exclusion Criteria:

* Known hypersensitivity to rhG-CSF or PEG-rhG-CSF;
* Female patients during pregnancy or lactation;
* The previous malignant tumors were not cured;
* Received chemotherapy or radiotherapy within 4 weeks before screening;
* Received PEG-rhG-CSF within 6 weeks before screening;
* Suffering from uncontrollable infectious diseases within 2 weeks before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2024-09-19 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of febrile neutropenia for chemotherapy cycle 1. | 21 days (Cycle 1 of chemotherapy treatment)
  Febrile neutropenia is defined as single temperature: ≥38.3 °C orally（axillary 38.1°C） or ≥38.0 °C（axillary 37.8°C） over 2h; and neutropenia: <500 neutrophils/mcL.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China